CLINICAL TRIAL: NCT00274599
Title: A Prospective, Randomised, Open-Label, Blinded-Endpoint, Parallel Group, Multicentre, Forced-Titration, 14-Week Treatment Study Comparing MICARDIS® (Telmisartan 40-80-80 mg, QD) and ALTACE® (Ramipril 2.5-5-10 mg, QD) in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring
Brief Title: PROBE Investigation of the Safety & Efficacy of Telmisartan (Micardis®) vs Ramipril (Altace®) Using ABPM in HTN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.392
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Ramipril

INTERVENTIONS:
Drug: Telmisartan
Drug: Ramipril

SUMMARY:
Demonstrate that telmisartan 80mg was at least as effective and possibly superior to ramipril 5mg & 10mg in lowering mean ambulatory DBP and SBP during the last 6 hrs of the 24-hr dosing interval in mild-to-moderate hypertensives at the end of 8 and 14 week treatment phases.

ELIGIBILITY:
Inclusion criteria:

* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP) and local legislation.
* Mild-to-moderate hypertension defined as a mean seated diastolic blood pressure of ≥95 mmHg and ≤109 mmHg, measured by manual cuff sphygmomanometer at Visit 2.
* Age 18 years or older (or 19 years if dictated by local State/Province policies).
* Ability to stop any current antihypertensive therapy without risk to the patient (investigator's discretion).
* 24-hour mean DBP of ≥85 mmHg at Visit 3 as measured by Ambulatory Blood Pressure Monitoring (ABPM).

Exclusion criteria:

* Pre-menopausal women (last menstruation ≤1 year prior to signing informed consent) who:

  * were not surgically sterile; or
  * were nursing, or
  * were of childbearing potential and were NOT practicing acceptable methods of birth control, or did NOT plan to continue practicing an acceptable method throughout the study. Acceptable methods of birth control included IUD, oral, implantable or injectable contraceptives. No exceptions were made.
* Night shift workers who routinely slept during the daytime and whose work hours included midnight to 4:00 a.m.
* Mean seated SBP ≥180 mmHg or mean seated DBP ≥110 mmHg during any visit of the placebo run-in period.
* Known or suspected secondary hypertension (e.g., phaeochromocytoma).
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters:
* Serum Glutamate-Oxaloacetate-Transaminase (Aspartate Aminotransferase) (SGOT (AST)) or Serum Glutamate-Pyruvate-Transaminase (Alanine Aminotransferase) (SGPT (ALT)) >2 times the upper limit of normal range, or
* Serum creatinine >2.3 mg/dL (or >203 μmol/l).
* Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney.
* Clinically relevant sodium depletion, hypokalaemia or hyperkalaemia.
* Uncorrected volume depletion.
* Further exclusion criteria apply

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2002-10-09 (Actual); Primary Completion 2003-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the last 6-hr mean DBP & SBP as measured by ABPM at the end of and 8-wk treatment period (T80 vs R5 mg) and 14-wk treatment period (T80 vs R10 mg) | Up to week 14

SECONDARY OUTCOMES:
Change from baseline in last 6-hr ABPM mean for: pulse pressure; DBP, SBP and PP; DBP/SBP/PP in the morning, daytime and nighttime periods of the 24-hr dosing interval; Change from baseline in mean, seated, trough DBP & SBP measured by manual cuff | Up to week 14

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (74):
- United States (43):
  - Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - Harold B. Betton, M.D., Little Rock, Arkansas
  - Attn: Ginger Paselk, Long Beach, California
  - Boehringer Ingelheim Investigational Site, Los Angeles, California
  - Boehringer Ingelheim Investigational Site, Orange, California
  - Boehringer Ingelheim Investigational Site, San Diego, California
  - Boehringer Ingelheim Investigational Site, Santa Ana, California
  - Boehringer Ingelheim Investigational Site, Santa Rosa, California
  - Boehringer Ingelheim Investigational Site, Vista, California
  - Boehringer Ingelheim Investigational Site, Hamden, Connecticut
  - Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - Boehringer Ingelheim Investigational Site, Boise, Idaho
  - Boehringer Ingelheim Investigational Site, Meridian, Idaho
  - Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - Boehringer Ingelheim Investigational Site, Orland Park, Illinois
  - GFI Pharmaceuticals, Evansville, Indiana
  - Boehringer Ingelheim Investigational Site, Newton, Kansas
  - Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - Boehringer Ingelheim Investigational Site, Metairie, Louisiana
  - Boehringer Ingelheim Investigational Site, Auburn, Maine
  - Boehringer Ingelheim Investigational Site, Moorestown, New Jersey
  - Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - Boehringer Ingelheim Investigational Site, East Syracuse, New York
  - Boehringer Ingelheim Investigational Site, White Plains, New York
  - Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - Boehringer Ingelheim Investigational Site, Portland, Oregon
  - Boehringer Ingelheim Investigational Site, Levittown, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Boehringer Ingelheim Investigational Site, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - Boehringer Ingelheim Investigational Site, Lacey, Washington
  - Boehringer Ingelheim Investigational Site, Lakewood, Washington
  - Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - Boehringer Ingelheim Investigational Site, Charleston, West Virginia
- Canada (31):
  - Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - Boehringer Ingelheim Investigational Site, Conquitlam, British Columbia
  - Boehringer Ingelheim Investigational Site, Riverview, New Brunswick
  - Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - Boehringer Ingelheim Investigational Site, Bay Roberts, Newfoundland and Labrador
  - Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - Boehringer Ingelheim Investigational Site, Exeter, Ontario
  - Boehringer Ingelheim Investigational Site, Hastings, Ontario
  - Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - Boehringer Ingelheim Investigational Site, London, Ontario
  - Boehringer Ingelheim Investigational Site, North York, Ontario
  - Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - Boehringer Ingelheim Investigational Site, Orléans, Ontario
  - 205-13085 Yonge St, Richmond Hill, Ontario
  - 155 Ontario Street, St. Catharines, Ontario
  - Boehringer Ingelheim Investigational Site, Thunder Bay, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Weston, Ontario
  - Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - Boehringer Ingelheim Investigational Site, Winnipeg, Ontario
  - Boehringer Ingelheim Investigational Site, Charlottetown, Prince Edward Island
  - 4 rue Robinson Nord, Granby, Quebec
  - Boehringer Ingelheim Investigational Site, Longueuil, Quebec
  - Boehringer Ingelheim Investigational Site, Pointe-Claire, Quebec
  - Boehringer Ingelheim Investigational Site, Saint-Léonard, Quebec
  - 725 6E Rue, Val-d'Or, Quebec
  - Boehringer Ingelheim Investigational Site, Regina, Saskatchewan
  - Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan